CLINICAL TRIAL: NCT07058064
Title: WATCH (Wearable Artificial inTelligence for Cardiac Function and Health Monitoring)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joerg Herrmann, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 25-002911; NCI-2025-04631 (Other: CTRP (Clinical Trial Reporting Program)); 25-002911 (Other: Mayo Clinic Institutional Review Board); HT94252510309 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Lymphoma; Sarcoma
MeSH Terms: conditions — Lymphoma; Sarcoma | interventions — Caves; Blood Specimen Collection; Surveys and Questionnaires; Clostridium perfringens epsilon-toxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cross-sectional Arm (Active Comparator): Lymphoma and sarcoma cancer survivors will be seen at one time point, 1 year after completion of anthracycline-based therapy.
  Interventions: Procedure: Electrocardiogram; Procedure: Echocardiogram; Procedure: LVEF echocardiogram; Procedure: Biospecimen collection; Other: Questionnaires
- Longitudinal Arm (Experimental): Lymphoma and sarcoma cancer survivors will be seen before the start of anthracycline-based therapy and followed every three months up to 1 year after completion of therapy. Longitudinal participants will have the option of recording ECG and cardio fitness data through an Apple Watch from before up to 1 year post anthracycline treatment.
  Interventions: Procedure: Electrocardiogram; Procedure: Echocardiogram; Procedure: LVEF echocardiogram; Other: Apple Watch; Procedure: Biospecimen collection; Other: Questionnaires; Other: Cardio-pulmonary exercise test; Other: 6 minute walk test; Other: Grip strength test

INTERVENTIONS:
Procedure: Electrocardiogram — All participants receive a standard 12-lead ECG when they present for follow-up 1 year after completion of anthracycline-based therapy. All participants will also record a 6-lead Kardia (AliveCor, Mountain View, CA, USA) and 1-lead Apple Watch (Apple, Cupertino, CA, USA) ECG with Mayo-owned or participant-owned devices.
  Longitudinal participants will receive an Apple Watch to use during this study if they do not have their own (and agree to download the app) and will be able to transmit ECGs anytime anywhere from their Apple Watch from before the initiation, all through the treatment, up to 1-year after anthracycline-based therapy. For validation, these participants will transmit ECGs from their smart watch at the time of routine follow-up visits (at 3-, 6- & 9-months post therapy visits) along with 6-lead Kardia ECGs, and 12-lead standard ECGs.
  Other Names: ECG; EKG
Procedure: Echocardiogram — All participants will have an echocardiogram as part of standard of care when they present for their follow-up 1 year after completion of anthracycline-based therapy.
  Other Names: echo; cardiac ultrasound; heart ultrasound
Procedure: LVEF echocardiogram — Participants will undergo a limited LVEF echocardiogram at the 6-month post therapy visit.
  Other Names: Left ventricular ejection fraction (LVEF) echocardiogram; LVEF echo
Other: Apple Watch — Longitudinal participants will receive an Apple Watch to use during this study if they do not have their own (and agree to download the app) and will be able to transmit ECGs anytime anywhere from their Apple Watch from before the initiation, all through the treatment, up to 1-year after anthracycline-based therapy. For validation, these participants will transmit ECGs from their smart watch at the time of routine follow-up visits (at 3-, 6- & 9-months post therapy visits) along with 6-lead Kardia ECGs, and 12-lead standard ECGs.
  Longitudinal participants will be asked to transmit weekly cardio fitness (estimates of peak VO2) from baseline to 1-year post therapy.
  Arms: Longitudinal Arm
Procedure: Biospecimen collection — Undergo blood draw
  Other Names: Blood draw
Other: Questionnaires — Participants fill out 2 questionnaires: 1) the Kansas City Cardiomyopathy-12 (KCCQ-12) Questionnaire, and 2) the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) ore 30 (EORTC QLQ-C30) to evaluate health related quality of life and heart failure symptoms.
Other: Cardio-pulmonary exercise test — Undergo CPET to assess the response of heart and lungs to exercise.
  Other Names: CPET
  Arms: Longitudinal Arm
Other: 6 minute walk test — Complete a 6MWT, to see how far participants can walk on a hard, flat surface for 6 minutes
  Other Names: 6MWT
  Arms: Longitudinal Arm
Other: Grip strength test — A hand-held device called a dynamometer will be used to measure the muscle strength in hand/forearm
  Arms: Longitudinal Arm

SUMMARY:
The purpose of this study is to find a cost effective cardiovascular (CV) surveillance of cancer survivors over long periods of time to prevent the risk of progression of heart failure (HF) and related morbidity and mortality. Mobile device-based artificial intelligence (AI)-electrocardiogram (ECG) can reliably detect cardiac dysfunction in lymphoma and sarcoma survivors and smart watch based surveillance for cardiotoxicity is feasible and reliable.

ELIGIBILITY:
Inclusion Criteria:

* ability to understand study procedures and being willing to comply with them for the entire study length
* diagnosis of lymphoma or sarcoma with new start or 1 year after completion of anthracycline therapy

Exclusion Criteria:

* LVEF <50% at baseline, or prior confirmed history of heart failure, persistent atrial fibrillation, left bundle branch block, or paced rhythm
* Unwilling or unable to give written informed consent
* Participants who have opted out of the Minnesota Research Authorization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2029-06-29 (Estimated); Study Completion 2029-06-29 (Estimated)

PRIMARY OUTCOMES:
Detection of left left ventricular ejection fraction (LVEF) <50% by AI-ECG | Baseline to 1 year follow-up
  Mobile device ECGs will be compared to standard 12-lead clinic ECGs for the AI algorithm to predict a reduced EF (EF <50%).
Change in AI-ECG based probability of an LVEF <50% using mobile device ECGs | Baseline to 1 year follow-up
  The change in probability of abnormal LVEF by AI-ECG using mobile device ECG will be compared between patients who do develop a reduction in LVEF over time versus those who do not.
Change in peak VO2 | Baseline to 1 year follow-up
  Volume of Oxygen (VO2) will be estimated by the Apple Watch algorithm (developed by Apple Inc.) and reviewed for change from baseline to 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Herrmann, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials